CLINICAL TRIAL: NCT02893800
Title: Assistive Technology for Dementia: Validation and Optimization of the Individual Benefits of Locating Systems in Dementia Care (VODINO)
Brief Title: Validation and Optimization of the Individual Benefits of Locating Systems in Dementia Care
Acronym: VODINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Alzheimer Society (Other)
Responsible Party: Principal Investigator, Oliver Peters, MD, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: VODINO_EA4/033/16
Record Dates: First submitted 2016-08-29; First posted 2016-09-09 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Dementia
Keywords: assistive technology; dementia care; tracking technology; locating systems; user experience
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Himatic locating system (Other): Locating system watch with GPS-technology (free available) Main functions: telephone function and location upon request via smartphone
  Interventions: Device: Locating system watch with GPS-technology
- ReSOS locating system (Other): Locating system watch with GPS-technology (free available) Main functions: telephone function and location upon request via smartphone
  Interventions: Device: Locating system watch with GPS-technology

INTERVENTIONS:
Device: Locating system watch with GPS-technology — Patients using locating system watches with embedded global positioning system (GPS) technology and telephone function; Caregivers using a Smartphone with an installed application to see the current location of the patient and with the possibility to call the patient

SUMMARY:
The project aims to make new technologies for locating people with dementia easier to use for the patients and those caring for them.

Objective: To systematically understand what improves the user experience of persons with dementia (PwD) and their primary caregivers (CG) with locating system watches to ultimately allow users to obtain more benefits from using these watches.

Aim: Improving the user experience of PwD and CG with locating system watches using a cross-over design and a theory-based educational session approach.

DETAILED DESCRIPTION:
This entire research field (assistive technology in dementia care) is based on the need to address care solutions for a growing number of PwD and CG in the absence of a cure for (Alzheimer's) dementia.

Methods: A user study with two free available locating watches. In educational sessions PwD obtain a locating watch and their CG a smartphone with the application of the locating watch installed on it. By using a cross-over design each dyad (PwD and CG) obtaining both locating systems. The designed educational session hopefully ease subsequent use and make it more enjoyable. The dyads will use each system over four weeks in their real environment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of all kinds of dementia or mild cognitive impairment

Exclusion Criteria:

* not able to move outside alone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Usability | 8 weeks
  ISONORM 9241/10 questionnaire (Prümper, 1997)

SECONDARY OUTCOMES:
Caregiver burden | 8 weeks
  Zarit Burden Interview (German version: Braun etal., 2010)
Acceptance and Practicability | 8 weeks
  Five-point likert scales and qualitative interview with open-ended questions
Subjective quality of life | 8 weeks
  European Health Interview Survey-Quality of Life (German version: Brähler et al., 2007)
Activities of Daily Living | 8 weeks
  BAYER-ADL (Hindmarch, 1998)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Peters, MD, Principal Investigator — Charité CBF
Locations (1):
- Charité University Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Aim: develop better business model designs to promote the adoption of assistive technologies in the field of dementia.
  In this context we share the qualitative data (transcripts of the interviews) with the department of business administration Prof.Dr.Wessel (Research Group "Health-IT and Business Model Innovation") of the Free University of Berlin.

REFERENCES:
- [Result] Megges H, Freiesleben SD, Rosch C, Knoll N, Wessel L, Peters O. User experience and clinical effectiveness with two wearable global positioning system devices in home dementia care. Alzheimers Dement (N Y). 2018 Nov 9;4:636-644. doi: 10.1016/j.trci.2018.10.002. eCollection 2018. PMID 30519629
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30519629/